CLINICAL TRIAL: NCT03879187
Title: Molecular and Hormonal Responses to Diet-Induced Insulin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Responsible Party: Principal Investigator, Carl Hulston, Senior Lecturer; Principal Investigator, Loughborough University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: R13-P171
Record Dates: First submitted 2019-03-12; First posted 2019-03-18 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Healthy
Keywords: High-fat diet; Insulin; Glucose; Muscle; eNOS; Isotopes
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Intervention Model Description: 15 healthy individuals were assessed before and after consuming a high-fat, high-energy diet for 7 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High-fat diet (Experimental): Participants underwent a 7 day high-fat, high-energy diet intervention with metabolic measurements before and after
  Interventions: Dietary Supplement: High-fat, high-energy diet

INTERVENTIONS:
Dietary Supplement: High-fat, high-energy diet — Participants consumed a diet that was high in fat and high in energy

SUMMARY:
This study determined the effect of 7 days of high-fat overfeeding on whole-body glycaemic control, glucose kinetics, skeletal muscle insulin signalling, and markers of skeletal muscle microvascular function in 15 healthy young individuals.

DETAILED DESCRIPTION:
Fifteen healthy, young individuals underwent metabolic testing before and after 7 days of high-fat overfeeding. We determined whole-body glycaemic control, glucose kinetics, skeletal muscle insulin signalling, and markers of skeletal muscle microvascular function. Stable isotope tracers were used to assess the rate of appearance of glucose from the gut, liver glucose output and whole-body glucose disposal. Insulin signalling was determined by Western blotting of skeletal muscle tissue. Microvascular function was assessed through the use of quantitative immunofluorescence microscopy. These measurements were performed both postabsorptively and following the ingestion of 50 grams of glucose + 15 grams of protein.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 40 years
* Physically active
* Non-smoker
* Not taking any medication known to interfere with the study
* No history of cardiovascular disease or diabetes
* Weight stable for the last 6 months

Exclusion Criteria:

* Outside of age range
* Sedentary
* Smoker
* Taking medication known to interfere with the study
* History of cardiovascular disease or diabetes
* Unstable weight within last 6 months

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2015-03-02 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2018-05-22 (Actual)

PRIMARY OUTCOMES:
Change in glucose concentration | Immediately before and after the 7 day high-fat diet (i.e., measurements were made 7 days apart)
  Venous blood samples were obtained the day before and the day after the 7 day high-fat diet. Glucose was reported as mmol/L.
Change in insulin concentration | Immediately before and after the 7 day high-fat diet (i.e., measurements were made 7 days apart)
  Venous blood samples were obtained the day before and the day after the 7 day high-fat diet. Insulin was reported as pmol/L.
Change in glucose kinetics (i.e., rate of appearance and disappearance) assessed using isotope tracers | Immediately before and after the 7 day high-fat diet (i.e., measurements were made 7 days apart)
  Glucose kinetics were assessed the day before and the day after the 7 day high-fat diet. Data expressed as umol/kg/min.
Change in skeletal muscle insulin signalling | Immediately before and after the 7 day high-fat diet (i.e., measurements were made 7 days apart)
  AKT and AS160 phosphorylation was determined by Western blotting of skeletal muscle. Data are expressed as arbitrary units.
Change in markers of microvascular function | Immediately before and after the 7 day high-fat diet (i.e., measurements were made 7 days apart)
  endothelial nitric oxide synthase was determined in terminal arterioles by quantitative immunofluorescence microscopy that was performed on sections of skeletal muscle tissue. Data presented as arbitrary units.

SECONDARY OUTCOMES:
Change intramuscular triglyceride content | Immediately before and after the 7 day high-fat diet (i.e., measurements were made 7 days apart)
  Intramuscular triglyceride content was determined by quantitative immunofluorescence microscopy that was performed on sections of skeletal muscle tissue. Data presented as arbitrary units.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parry SA, Turner MC, Woods RM, James LJ, Ferguson RA, Cocks M, Whytock KL, Strauss JA, Shepherd SO, Wagenmakers AJM, van Hall G, Hulston CJ. High-Fat Overfeeding Impairs Peripheral Glucose Metabolism and Muscle Microvascular eNOS Ser1177 Phosphorylation. J Clin Endocrinol Metab. 2020 Jan 1;105(1):dgz018. doi: 10.1210/clinem/dgz018. PMID 31513265